CLINICAL TRIAL: NCT01670916
Title: Probiotics to Prevent NEC Stage II+ in Very Preterm Infants - a Historical Control Study
Brief Title: Probiotics to Prevent NEC - a Historical Control Study
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gorm Greisen, professor, consultant neonatologist, Rigshospitalet, Denmark
Other Study IDs: RHNEO-NEC01
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing enterocolitis; Probiotics; Preterm; Infant
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth | interventions — Probiotics

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (2):
- Probiotics: Capsule with 1 x 10**9 Lactobacillus rhamnosus GG and 1 x 10**8 Bifidobacterium BB12. Two capsules once a day. The capsules are opened and the content is dissolved in mother's milk or water if the baby is given any milk. In tube fed infants, two drops are given in the mouth and the rest in the nasogastric tube.
  Interventions: Dietary Supplement: probiotics
- Control: Probiotics never given

INTERVENTIONS:
Dietary Supplement: probiotics — Capsule with 1 x 10**9 Lactobacillus rhamnosus GG and 1 x 10**8 Bifidobacterium BB12. Two capsules once a day. The capsules are opened and the content is dissolved in mother's milk or water if the baby is given any milk. In tube fed infants, two drops are given in the mouth and the rest in the nasogastric tube.
  Other Names: Bifiform, Ferrosan A/S; Idoform, Ferronan A/S
  Groups: Probiotics

SUMMARY:
Probiotics is given routinely to infants admitted to the department of neonatology during the first 3 days of life with gestational age less than 30 weeks since March 2010. The incidence of necrotizing enterocolitis Bell stage II and III will be assessed blindly from clinical records. It is hypothesised that the incidence of NEC will decrease. Infants admitted from 1 March 2010 to 28 February 2013 will be compared to infants admitted 1 Dec 2007 to 30 Nov 2009 will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 30 weeks
* Admission during the first 3 days of life

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants admitted for special or intensive care
Sampling Method: Non-Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
NEC | From birth until discharge home
  The clinical records of infants who had a discharge diagnosis of necrotizing enterocolitis are selected. Records of infants who had a prescription of metronidazole for a non-preventive purpose is added. The clinical records are abstracted. The abstracts and X-rays are presented to a review board that are blinded to the period of birth. The board classifies the cases as NEC-I, NEC-II, NEC-III, focal intestinal perforation, and OTHER.
  NEC-II/III is the primary outcome.

SECONDARY OUTCOMES:
Death with NEC | Birth to discharge home
  Death with a review board classification of NEC-II/III
Death | Birth to discharge home

OTHER OUTCOMES:
Positive culture of probiotic bacteria | Birth to discharge from Rigshospitalet
  Growth of lactobacilli or bifidobacteria from a normally sterile fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Lambaek ID, Fonnest G, Gormsen M, Brok J, Greisen G. Probiotics to prevent necrotising enterocolitis in very preterm infants. Dan Med J. 2016 Mar;63(3):A5203. PMID 26931192